CLINICAL TRIAL: NCT01993745
Title: The Analysis of Heart Rate Variability With 24hrs Holter ECG and Serum Cardiac Fibrosis Markers in Critical Illness Patients Who Are With Cardiogenic Shock, With ECMO or IABP Support, or With APACH II Score >25)
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200804046R
Record Dates: First submitted 2013-10-29; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Cardiogenic Shock,; With ECMO or IABP Support,; With APACH II Score >25)
Keywords: ECMO; APACH II score
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study group: ECMO Patients survived
- Control: ECMO Patient died

SUMMARY:
The study is to show the prognostic factor of HRV parameter and cardiac fibrosis markers in critical illness patients

DETAILED DESCRIPTION:
The analysis of Heart Rate Variability with 24hrs Holter ECG and serum cardiac fibrosis markers in critical illness patients who are with cardiogenic shock, with ECMO or IABP support, or with APACH II score >25)

ELIGIBILITY:
Inclusion Criteria:

* critical illness patients who are with cardiogenic shock, with ECMO or IABP support, or with APACH II score >25)

Exclusion Criteria:

* pacemaker rhythm, not sign the permit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult age>18 years old
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability and serum cardiac fibrosis markers in critical illness patients | 2-4weeks
  1. Outcome measurement:
     The measure is a composite outcome measure consisting of multiple measures (results to be reported as a single value for each Arm/Group), no changes are required
  2. List the primary condition or disease being studied Shock needing ECMO support

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan